CLINICAL TRIAL: NCT02597855
Title: Short-term Efficacy of Intravitreal Afilibercept Depending on Subtypes of Polypoidal Choroidal Vasculopathy: Polypoidal Choroidal Neovascularization or Idiopathic Choroidal Vasculopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Assistant Professor, Yeungnam University College of Medicine
Other Study IDs: YUMC2015-08-036
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 polypoidal choroidal vasculopathy: Monthly intravitreal aflibercept injection for 3 months and 1 additional injection after 2 months. Indocyanine green angiography was used to classify the type of PCV and evaluate the polyp closure rate.
  Interventions: Drug: Aflibercept; Drug: Indocyanine green angiography (intraveonus indocyanine green dye)
- Type 2 polypoidal choroidal vasculopathy: Monthly intravitreal aflibercept injection for 3 months and 1 additional injection after 2 months. Indocyanine green angiography was used to classify the type of PCV and evaluate the polyp closure rate.
  Interventions: Drug: Aflibercept; Drug: Indocyanine green angiography (intraveonus indocyanine green dye)

INTERVENTIONS:
Drug: Aflibercept — Total 4 times of intravitreal aflibercept injection was performed
  Other Names: Eylea
Drug: Indocyanine green angiography (intraveonus indocyanine green dye) — At initial visit, indocyanine green angiography was performed. After 1 month of third Aflibercept injection, indocyanine green angiography was performed to evaluate polyp closure.

SUMMARY:
To compare the short-term effect of intravitreal aflibercept injection between two subtypes of polypoidal choroidal vasculopathy

DETAILED DESCRIPTION:
The subjects were classified into two subtypes (type 1 and type 2 polypoidal choroidal vasculopathy) based on the presence or the absence of both of a feeder and a draining vessels on indocyanine green angiography. All received intravitreal injection of aflibercept (2.0 mg) at baseline and months 1, 2 and 4.

ELIGIBILITY:
Inclusion Criteria:

1. symptomatic typical PCV accompanying branch vascular network involving subfoveal area
2. signed informed consent; and
3. over 6 months follow-up period after enrollment.

Exclusion Criteria:

1. retinal diseases other than PCV
2. extrafoveal PCV not involving subfoveal area
3. massive subretinal hemorrhage blocking polypoidal lesion on ICGA
4. severe media opacity such as senile cataract
5. previous history of intravitreal injection
6. previous intraocular surgery history except cataract surgery which was done more than 3 months.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients were recruited from the retinal clinic of the Yeungnam university hospital. Recruitment started on October 01 2015 to March 31 2016.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University College of Medicine, Daegu, South Korea

REFERENCES:
- [Derived] Jeong S, Sagong M. Short-term efficacy of intravitreal aflibercept depending on angiographic classification of polypoidal choroidal vasculopathy. Br J Ophthalmol. 2017 Jun;101(6):758-763. doi: 10.1136/bjophthalmol-2016-309144. Epub 2016 Sep 5. PMID 27597740

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Type 1 Polypoidal Choroidal Vasculopathy | Type 2 Polypoidal Choroidal Vasculopathy
Started | 18 | 14
Completed | 16 | 13
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Type 1 Polypoidal Choroidal Vasculopathy; Type 2 Polypoidal Choroidal Vasculopathy: Monthly intravitreal aflibercept injection for 3 months and 1 additional injection after 2 months from third injection.
  At initial visit, indocyanine green angiography was performed. After 1 month of third Aflibercept injection, indocyanine green angiography was performed to evaluate polyp closure.
- Total: Total of all reporting groups
Arm/Group | Type 1 Polypoidal Choroidal Vasculopathy | Type 2 Polypoidal Choroidal Vasculopathy | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (7.4) | 64.2 (6.6) | 67.2 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Regression Rate of Polyp on Indocyanine Green Angiography
Description: Indocyanine green angiography performed initially and at 3 months were used to determine the polyp regression. The definition of complete polyp regression is that the polyps at initial visit disappeared at 3 months on indocyanine green angiography. The partial regression means the polyps remain, but the size decreased >30%.
Time Frame: 3 months
Population: Participants who were finished 6 months follow up period.
Measure: Number; unit: participants
Arm/Group | Type 1 Polypoidal Choroidal Vasculopathy | Type 2 Polypoidal Choroidal Vasculopathy
Number analyzed (Participants) | 16 | 13
participants
  Complete polyp regression | 13 | 4
  Partial polyp regression | 3 | 7
  No regression | 0 | 2
Statistical Analysis 1: Comparison: Type 1 Polypoidal Choroidal Vasculopathy vs Type 2 Polypoidal Choroidal Vasculopathy; The difference of polyp regression rate between two groups were compared; Test type: Superiority or Other; p < 0.05, Fisher Exact

2. Secondary Outcome: Best Corrected Visual Acuity
Description: Best corrected visual acuity assessed at baseline, 3 months, and 6 months
Time Frame: baseline, 3 months, and 6 monthsc
Population: Participants who were finished 6 months follow up period.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Type 1 Polypoidal Choroidal Vasculopathy | Type 2 Polypoidal Choroidal Vasculopathy
Number analyzed (Participants) | 16 | 13
LogMAR
  3 months | 0.39 (0.36) | 0.54 (0.34)
  6 months | 0.44 (0.26) | 0.49 (0.36)
  Baseline | 0.76 (0.41) | 0.62 (0.30)
Statistical Analysis 1: Comparison: Type 1 Polypoidal Choroidal Vasculopathy vs Type 2 Polypoidal Choroidal Vasculopathy; best corrected visual acuity was compared between two groups; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); The Mann-Whitney test was used for a comparison of best corrected visual acuity assessed at baseline, 3 months, and 6 months between type1 and type2

ADVERSE EVENTS:
Arm/Group | Type 1 Polypoidal Choroidal Vasculopathy | Type 2 Polypoidal Choroidal Vasculopathy
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 0/18 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No